CLINICAL TRIAL: NCT04878185
Title: Optimizing Physical Function Before Surgery: Effects on Complications and Physical Function After Gastrointestinal Cancer Surgery in Older People at Risk- A Randomized Controlled Trial
Brief Title: Optimizing Physical Function Before Cancer Surgery in Older People at Risk
Acronym: CanOptiPhys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Elisabeth Rydwik, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPN2015/1179-31
Record Dates: First submitted 2021-04-06; First posted 2021-05-07 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer; Postoperative Complications
Keywords: Preoperative Exercise
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): A high-intensity, home-based, exercise program consisting of inspiratory muscle training (IMT), endurance- and functional strength exercise. The sessions will supervised by a physiotherapist during six occasions and start 2-3 weeks before surgery. IMT will be conducted with an intensity starting from 50 % of maximal capacity, with a self-reported effort of 5-7 on the Borgs CR-10 scale. Endurance and functional strength exercises will be performed at a self-reported effort of 7-8. Interval training, chair stand- and step-up exercises will be key components of the exercise program. Furthermore, the program will include task-specific exercises based on the participants self-expressed needs.
  On non-supervised days, participants will perform IMT twice a day as well as endurance and strength training, 2-3 days per week with 1-2 days per week of active recovery in the form of moderate intensity walks. This will be monitored with an activity journal and an accelerometer.
  Interventions: Other: Exercise
- Control group (No Intervention): Participants in the control group receive pre- and postoperative care as usual. In addition, they will be encouraged to follow the WHO guidelines of moderate intensity aerobic physical activity for at least 150 min per week. Their activity level will be monitored with an accelerometer.

INTERVENTIONS:
Other: Exercise — Preoperative exercise
  Arms: Exercise

SUMMARY:
This randomized controlled trial is a multicentre study designed to explore the effects of preoperative exercise on physical fitness, postoperative complications, recovery, and health-related quality of life in older individuals at risk scheduled to undergo colorectal cancer surgery. The hypothesis is that older patients with low preoperative physical capacity will benefit from preoperative exercise in terms of lower risk for postoperative complications and improved recovery after surgery.

DETAILED DESCRIPTION:
Reduced physical capacity and performance associated with advancing age may decrease the ability to withstand the strain of a major surgical intervention. Exercise prior to surgery is a key component of prehabilitation. The goal of prehabilitation is to enhance preoperative physical fitness to attenuate postoperative decline and possibly decrease the risk of postoperative complications.

A previous observational study showed that better preoperative physical performance in measures of walking distance, leg strength, inspiratory muscle strength and maximal gait speed reduced the risk of severe postoperative complications for older patients undergoing abdominal cancer surgery. Furthermore, gait speed has been suggested to add information to current preoperative risk screening, where a cut of value of a maximal gait speed below 2 meters/second indicates a higher risk for postoperative complications.

This planned trial will be conducted in cooperation with the Karolinska University Hospital, Ersta Hospital, The Stockholm South General Hospital and several primary care units in Stockholm. To target older patients at risk, patients aged 65 and older with a maximal gait speed under 2 meters/second will be included. Participants will be randomized to either intervention- or control group and trained physiotherapists or nurses from the hospitals, will conduct the assessments. All baseline measures will be collected before randomization.

The implementation of standardized cancer care pathways in Sweden has led to reduced time between diagnosis to curative treatment. For colorectal surgery, the time from decision to treatment is set to two weeks. Therefore, an exercise program aimed to enhance physical function prior to surgery require a high intensity and high frequency approach. The exercise program will be home-based and consist of inspiratory muscle training, endurance- and strength exercise under the supervision of trained physiotherapists from primary care units. To assess feasibility of the planned intervention, a pilot study was conducted. The results showed high compliance and acceptability among the participants which provides a starting point for this larger study designed to explore the effects of preoperative exercise on:

1. Preoperative physical function in a short-term perspective
2. Postoperative complications and functional decline
3. Length of in-hospital stay, mortality, health-related quality of life, physical activity level and independency in activities in daily living in a long-term perspective

ELIGIBILITY:
Inclusion Criteria:

* Scheduled surgery due to colorectal cancer or liver metastases from colorectal cancer
* Age ≥65
* A maximal walking speed below 2 meters per second
* Understands and speaks the Swedish language

Exclusion Criteria:

* Planned hyperthermic intraperitoneal chemotherapy (HIPEC) procedure or flap surgery
* Health conditions that prevent participation in assessment or exercise. Such conditions include, but are not limited to, unstable heart disease, severe systematic illness or orthopaedic conditions that may prohibit exercise.
* The need for surgery within 2 weeks
* Permanent wheelchair user
* Residence outside of Stockholm County

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Postoperative Complications 30 days post-surgery | 30 days post-surgery
  The Clavien-Dindo classification system will be used to describe the occurence of post-operative complications.
Change in maximal walking distance | Baseline, completion immediately after intervention, and day of hospital discharge (average: 5 days)
  The 6-minute walk test will be used to assess physical endurance. The test requires subjects to walk as far as possible during 6 minutes. Outcome is metres walked.

SECONDARY OUTCOMES:
Length of hospital stay | Baseline (day of hospital admission), day of hospital discharge (average: 5 days)
  The number of days spent at hospital. Data will be collected from the medical records. Outcome is number of days.
Quality of life as assessed by the EORTC QLQ-C30 | Baseline, 6 and 12 months post-surgery
  The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire core-30 (EORTC QLQ-C30) and the supplemental Elderly Cancer Patients Module will be used to assess quality of life. The scale is comprised of nine subscales: one global health status scale, five functioning scales and three symptom scales. The scales range from 0-100 scores. Higher scores for the global health status scale and functioning scales indicate better outcomes. For the symptom scales, higher scores indicate worse outcomes.
Quality of life as assessed by the EORTC QLQ-ELD14 | Baseline, 6 and 12 months post-surgery
  The European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire for the Elderly Cancer Patients Module (EORTC QLQ-ELD14) will be used to assess quality of life. The scale is comprised of five subscales: mobility, family support, worries about the future, maintaining autonomy and purpose, and burden of illness. The scales range from 0-100 scores. For the family support scale and the autonomy and purpose scale, higher scores indicate better outcomes. For the mobility, worries and burden of illness scales, higher scores indicate worse outcomes.
Destination of discharge from the hospital | Day of hospital discharge (average: 5 days)
  Data on destination of discharge will be collected from the medical journal. The information will be categorized into home, rehabilitation facility or further care (in e.g a geriatric clinic or residential care).
Patient-reported symptoms | 2-3 days post-surgery, day of hospital discharge (average: 5 days), and 6 months post-surgery
  The Postoperative Recovery Profile. The scale consists of physical symptoms, physical function, psychological and social impact and activity. The results are divided in 5 categories from not recovered at all to fully recovered.
Delirium | 2-3 days post-surgery
  Confusion Assessment Method consists of 9 item, if you fulfill one of the items 1-4, you are diagnosed with confusion.
Change in lower extremity strength | Baseline, completion immediately after intervention, and day of hospital discharge (average: 5 days)
  The 30-second chair stand test will be used to measure functional lower extremity strength. Outcome is the number of times the patient comes to a full standing position in 30 seconds.
Change in maximal inspiratory muscle strength | Baseline, completion immediately after intervention, and day of hospital discharge (average: 5 days)
  Micro respiratory pressure meter is measured using the MicroRPM.
Level of independence in daily living | Baseline, 6 and 12 months post-surgery
  The ADL-staircase is an hierarchical scale with 10 items including both personal and instrumental activities ranging from inpedendent to dependent.
Physical activity level | Baseline, 6 and 12 months post-surgery
  Physical Activity Scale for the Elderly includes time spent in sitting, exercise, leisure, household/gardening and work/voluntary activities. It scores from 0 to 400, higher score indicate higher activity level.
Mortality | Baseline (post-surgery), 12, 24, and 36 months post-surgery
  Mortality data will be collected from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Rydwik, Assoc prof, Principal Investigator — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Karolinska University Hospital Huddinge, Huddinge, Karolinska Institutet
  - Karolinska University Hospital Solna, Stockholm
  - Ersta hospital, Stockholm
  - Stockholm South General Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Data is not publicly available, but available upon request.
Supporting Information: Study Protocol
Time Frame: After study completion 2024
Access Criteria: Requests for access to the data can be put to our Research Data Office (rdo@ki.se) at Karolinska Institutet, and will be handled according to the relevant legislation. This will require a data processing agreement or similar with the recipient of the data.

REFERENCES:
- [Background] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Background] Topp R, Ditmyer M, King K, Doherty K, Hornyak J 3rd. The effect of bed rest and potential of prehabilitation on patients in the intensive care unit. AACN Clin Issues. 2002 May;13(2):263-76. doi: 10.1097/00044067-200205000-00011. PMID 12011598
- [Background] Karlsson E, Egenvall M, Farahnak P, Bergenmar M, Nygren-Bonnier M, Franzen E, Rydwik E. Better preoperative physical performance reduces the odds of complication severity and discharge to care facility after abdominal cancer resection in people over the age of 70 - A prospective cohort study. Eur J Surg Oncol. 2018 Nov;44(11):1760-1767. doi: 10.1016/j.ejso.2018.08.011. Epub 2018 Aug 29. PMID 30201418
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Katsura M, Kuriyama A, Takeshima T, Fukuhara S, Furukawa TA. Preoperative inspiratory muscle training for postoperative pulmonary complications in adults undergoing cardiac and major abdominal surgery. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD010356. doi: 10.1002/14651858.CD010356.pub2. PMID 26436600
- [Derived] Danielsson J, Engstrom Sid J, Andersson M, Nygren-Bonnier M, Egenvall M, Hagstromer M, Vossen LE, Dohrn IM, Rydwik E. Optimizing Physical Fitness Before Colorectal Cancer Surgery (CANOPTIPHYS): The Effect of Preoperative Exercise on Pre- and Postoperative Physical Fitness in Older people - A Randomized Controlled Trial. J Prim Care Community Health. 2025 Jan-Dec;16:21501319251346417. doi: 10.1177/21501319251346417. Epub 2025 Jun 17. PMID 40525350
- [Derived] Andersson M, Egenvall M, Danielsson J, Thorell A, Sturesson C, Soop M, Nygren-Bonnier M, Rydwik E. CANOPTIPHYS study protocol: Optimising PHYSical function before CANcer surgery: effects of pre-operative optimisation on complications and physical function after gastrointestinal cancer surgery in older people at risk-a multicentre, randomised, parallel-group study. Trials. 2023 Jan 19;24(1):41. doi: 10.1186/s13063-022-07026-w. PMID 36658653